CLINICAL TRIAL: NCT03519256
Title: A Phase 2, Randomized, Open-label Study of Nivolumab or Nivolumab/BMS-986205 Alone or Combined With Intravesical BCG in Participants With BCG-Unresponsive, High-Risk, Non-Muscle Invasive Bladder Cancer
Brief Title: A Study of Nivolumab or Nivolumab Plus Experimental Medication BMS-986205 With or Without Bacillus Calumette-Guerin (BCG) in BCG Unresponsive Bladder Cancer That Has Not Invaded Into the Muscle Wall of the Bladder
Acronym: CheckMate 9UT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient Enrollment
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-9UT; 2017-003581-27 (EudraCT Number)
Record Dates: First submitted 2018-04-17; First posted 2018-05-08 (Actual); Results first posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Urinary Bladder Neoplasms
Keywords: Bladder Cancer; BCG-unresponsive; Nivolumab; Intravesical BCG; NMIBC; Non-Muscle Invasive; BMS-986205; CheckMate 9UT
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — Nivolumab; linrodostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Nivolumab monotherapy (Experimental)
  Interventions: Biological: Nivolumab
- Nivolumab + BCG (Experimental)
  Interventions: Biological: Nivolumab; Biological: BCG
- Nivolumab + BMS-986205 (Experimental)
  Interventions: Biological: Nivolumab; Drug: BMS-986205
- Nivolumab + BMS-986205 + BCG (Experimental)
  Interventions: Biological: Nivolumab; Biological: BCG; Drug: BMS-986205

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
Biological: BCG — Specified dose on specified days
  Other Names: Bacillus Calumette-Guerin
  Arms: Nivolumab + BCG; Nivolumab + BMS-986205 + BCG
Drug: BMS-986205 — Specified dose on specified days
  Arms: Nivolumab + BMS-986205; Nivolumab + BMS-986205 + BCG

SUMMARY:
A study to evaluate the safety and tolerability of nivolumab or nivolumab Plus BMS-986205 with or without BCG in BCG-Unresponsive non-muscle invasive Bladder Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically demonstrated BCG-unresponsive, carcinoma in situ (CIS)-containing high-risk non-muscle-invasive bladder cancer (NMIBC) defined as CIS with or without papillary component
* Participants must have CIS to be eligible.
* Predominant histologic component (> 50%) must be urothelial (transitional cell) carcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1

Exclusion Criteria:

* Sign of locally advanced disease or metastatic bladder cancer
* Urothelial cancer (UC) in the upper genitourinary tract (kidneys, renal collecting systems, ureters) within 24 months of enrollment
* Prior immuno-oncology therapy

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (88):
- United States (25):
  - Local Institution - 0044, Los Angeles, California
  - Local Institution - 0081, Riverside, California
  - Local Institution - 0087, San Francisco, California
  - Local Institution - 0125, Tampa, Florida
  - Local Institution - 0056, Hapeville, Georgia
  - Local Institution - 0023, New Lenox, Illinois
  - Wichita Urology Group, Wichita, Kansas
  - Local Institution - 0001, Baltimore, Maryland
  - Local Institution - 0077, Ann Arbor, Michigan
  - Local Institution - 0032, Minneapolis, Minnesota
  - Local Institution - 0040, Omaha, Nebraska
  - Local Institution - 0144, New Brunswick, New Jersey
  - Deleware Valley Urology, LLC, Voorhees Township, New Jersey
  - Local Institution - 0051, New York, New York
  - Local Institution - 0058, Columbus, Ohio
  - Local Institution - 0036, Bala-Cynwyd, Pennsylvania
  - Local Institution - 0049, Charleston, South Carolina
  - Local Institution - 0002, Myrtle Beach, South Carolina
  - Local Institution - 0057, Chattanooga, Tennessee
  - Urology Clinics Of North Texas, Pa, Dallas, Texas
  - Local Institution - 0048, Houston, Texas
  - Local Institution - 0140, Houston, Texas
  - Local Institution - 0047, Lubbock, Texas
  - Urology San Antonio Research, Pa, San Antonio, Texas
  - Local Institution - 0141, Seattle, Washington
- Argentina (6):
  - Local Institution - 0068, Capital Federal, Buenos Aires
  - Local Institution - 0065, Capital Federal, Distrito Federal
  - Local Institution - 0089, Ciudad Autonoma Buenos Aires, Distrito Federal
  - Local Institution, Viedma, Río Negro Province
  - Instituto Oncologico De Cordoba, Córdoba
  - Local Institution - 0137, Mendoza
- Australia (2):
  - Local Institution - 0146, Camperdown, New South Wales
  - Local Institution - 0148, St Leonards, New South Wales
- Brazil (7):
  - Local Institution - 0072, Fortaleza, Ceará
  - Local Institution - 0151, Curitiba, Paraná
  - Local Institution - 0073, Porto Alegre, Rio Grande do Sul
  - Local Institution, Itacorubi, Florianopolis, Santa Catarina
  - Local Institution - 0078, Jaú, São Paulo
  - Local Institution - 0150, Rio de Janeiro
  - Local Institution - 0074, São Paulo
- Canada (4):
  - Local Institution - 0143, North York, Ontario
  - Local Institution - 0086, Toronto, Ontario
  - Local Institution - 0084, Toronto, Ontario
  - Local Institution - 0046, Québec, Quebec
- Chile (2):
  - Local Institution - 0154, Santiago, Santiago Metropolitan
  - Local Institution - 0069, Santiago, Santiago Metropolitan
- China (17):
  - Local Institution - 0128, Beijing, Beijing Municipality
  - Local Institution - 0131, Beijing, Beijing Municipality
  - Local Institution - 0116, Beijing, Beijing Municipality
  - Local Institution - 0099, Beijing, Beijing Municipality
  - Local Institution - 0129, Chongqing, Chongqing Municipality
  - Local Institution - 0108, Fuzhou, Fujian
  - Local Institution - 0117, Guangzhou, Guangdong
  - Local Institution - 0102, Nanjing, Jiangsu
  - Local Institution - 0109, Nanchang, Jiangxi
  - Local Institution - 0112, Jinan, Shandong
  - Local Institution - 0111, Yantai, Shandong
  - Local Institution - 0098, Shanghai, Shanghai Municipality
  - Local Institution - 0094, Shanghai, Shanghai Municipality
  - Local Institution - 0097, Shanghai, Shanghai Municipality
  - Local Institution - 0120, Chengdu, Sichuan
  - Local Institution - 0133, Tianjin, Tianjin Municipality
  - Local Institution - 0126, Hangzhou, Zhejiang
- France (5):
  - Local Institution - 0027, Suresnes, Hauts-de-Seine
  - Local Institution - 0028, Angers, Maine-et-Loire
  - Local Institution - 0031, Bordeaux
  - Local Institution - 0088, Lille
  - Local Institution - 0091, Strasbourg
- Local Institution - 0093, Hong Kong, Hong Kong
- Italy (3):
  - IRCCS Istituto Nazionale Tumori Milano, Milan
  - Instituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Azienda Ospedaliera Universitaria Pisana, Pisa
- Mexico (2):
  - Local Institution - 0062, Tuxtla Gutiérrez, Chiapas
  - Local Institution - 0055, Mexico City, Mexico City
- Netherlands (3):
  - Local Institution - 0004, Amsterdam
  - Local Institution - 0003, Nijmegen
  - Local Institution - 0005, Utrecht
- Russia (3):
  - Local Institution - 0070, Omsk
  - Local Institution - 0054, Saint Petersburg
  - Local Institution - 0153, Saint Petersburg
- Spain (4):
  - Local Institution, Madrid
  - Local Institution - 0033, Málaga
  - Local Institution - 0139, Santander
  - Local Institution - 0136, Valencia
- United Kingdom (4):
  - Local Institution, Chelmsford, Essex
  - Local Institution, London, Greater London
  - Local Institution - 0013, Southampton, Hampshire
  - Local Institution - 0015, Lancaster

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A safety lead-in was conducted in participants randomized to receive bacillus Calmette-Guerin (BCG) and nivolumab without BMS-986205 (Arm B), and Nivolumab Plus BMS-986205 Plus Intravesical BCG (Arm D) to determine safe-dose levels to be administered during the treatment phase.
Groups:
- Arm A: Nivolumab: Nivolumab 480 mg IV every 4 weeks (Q4W) for up to 52 weeks (12 months).
- Arm B: Nivolumab Plus Intravesical BCG: Nivolumab 480 mg IV every 4 weeks (Q4W) for up to 52 weeks (12 months) and intravesical BCG (induction) weekly for 6 weeks followed by maintenance intravesical BCG weekly for 3 weeks at 3 months, 6 months and 12 months following the first intravesical dose.
- Arm C: Nivolumab Plus BMS-986205: Nivolumab 480 mg IV every 4 weeks (Q4W) and 100 mg oral BMS-986205 daily for up to 52 weeks (12 months).
- Arm D: Nivolumab Plus BMS-986205 Plus Intravesical BCG: Nivolumab 480 mg IV every 4 weeks (Q4W), 100 mg oral BMS-986205 daily for up to 52 weeks (12 months), and intravesical BCG (induction) weekly for 6 weeks followed by maintenance intravesical BCG weekly for 3 weeks at 3 months, 6 months, and 12 months following the first intravesical dose.
Period: Overall Study
Arm/Group | Arm A: Nivolumab | Arm B: Nivolumab Plus Intravesical BCG | Arm C: Nivolumab Plus BMS-986205 | Arm D: Nivolumab Plus BMS-986205 Plus Intravesical BCG
Started | 16 | 26 | 17 | 10
Safety-Lead In Phase | 0 | 10 | 0 | 10
Completed | 6 | 15 | 2 | 3
Not Completed | 10 | 11 | 15 | 7
Not completed — Disease recurrence | 4 | 4 | 5 | 2
Not completed — Study drug toxicity | 0 | 2 | 5 | 2
Not completed — Adverse event unrelated to study drug | 0 | 1 | 1 | 0
Not completed — Participant request to discontinue study treatment | 0 | 0 | 0 | 2
Not completed — Other reasons | 0 | 0 | 2 | 0
Not completed — Disease progression | 6 | 3 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Nivolumab | Arm B: Nivolumab Plus Intravesical BCG | Arm C: Nivolumab Plus BMS-986205 | Arm D: Nivolumab Plus BMS-986205 Plus Intravesical BCG | Total
Number analyzed (Participants) | 16 | 26 | 17 | 10 | 69
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.8 (11.1) | 69.0 (9.4) | 69.1 (12.3) | 69.9 (16.4) | 67.5 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 5 | 1 | 12
  Male | 14 | 22 | 12 | 9 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 3 | 1 | 6
  Not Hispanic or Latino | 11 | 23 | 8 | 9 | 51
  Unknown or Not Reported | 5 | 1 | 6 | 0 | 12
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 13 | 26 | 17 | 10 | 66
  Asian | 3 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. AEs are reported using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: From first dose to 30 days post last dose of study treatment (an average of 45 weeks up to approximately 64 weeks)
Population: All randomized participants who received at least one dose of any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab | Arm B: Nivolumab Plus Intravesical BCG | Arm C: Nivolumab Plus BMS-986205 | Arm D: Nivolumab Plus BMS-986205 Plus Intravesical BCG
Number analyzed (Participants) | 16 | 26 | 17 | 10
Participants | 15 | 26 | 15 | 10

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose:
  * Results in death
  * Is life-threatening (an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe)
  * Requires inpatient hospitalization or causes prolongation of existing hospitalization.
  SAEs are reported using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: From first dose to 30 days post last dose of study treatment (an average of 45 weeks up to approximately 64 weeks)
Population: All randomized participants who received at least one dose of any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab | Arm B: Nivolumab Plus Intravesical BCG | Arm C: Nivolumab Plus BMS-986205 | Arm D: Nivolumab Plus BMS-986205 Plus Intravesical BCG
Number analyzed (Participants) | 16 | 26 | 17 | 10
Participants | 2 | 4 | 6 | 4

3. Primary Outcome: Number of Participants With Adverse Events (AEs) Leading to Discontinuation of Study Treatment
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. AEs leading to discontinuation are reported using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: From first dose to 30 days post last dose of study treatment (an average of 45 weeks up to approximately 64 weeks)
Population: All randomized participants who received at least one dose of any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab | Arm B: Nivolumab Plus Intravesical BCG | Arm C: Nivolumab Plus BMS-986205 | Arm D: Nivolumab Plus BMS-986205 Plus Intravesical BCG
Number analyzed (Participants) | 16 | 26 | 17 | 10
Participants | 1 | 4 | 8 | 7

4. Primary Outcome: Number of Participants Immune-Mediated Adverse Events (IMAEs)
Description: IMAEs are AEs consistent with an immune-mediated mechanism or immune-mediated component for which non-inflammatory etiologies (eg, infection or tumor progression) have been ruled out. IMAEs can include events with an alternate etiology which were exacerbated by the induction of autoimmunity IMAEs are reported using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: From first dose to 30 days post last dose of study treatment (an average of 45 weeks up to approximately 64 weeks)
Population: All randomized participants who received at least one dose of any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab | Arm B: Nivolumab Plus Intravesical BCG | Arm C: Nivolumab Plus BMS-986205 | Arm D: Nivolumab Plus BMS-986205 Plus Intravesical BCG
Number analyzed (Participants) | 16 | 26 | 17 | 10
Participants | 1 | 10 | 6 | 5

5. Primary Outcome: Number of Participants Who Died
Description: Number of participants who died.
Time Frame: From first dose to 100 days post last dose of study treatment (an average of 45 weeks up to approximately 74 weeks)
Population: All randomized participants who received at least one dose of any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab | Arm B: Nivolumab Plus Intravesical BCG | Arm C: Nivolumab Plus BMS-986205 | Arm D: Nivolumab Plus BMS-986205 Plus Intravesical BCG
Number analyzed (Participants) | 16 | 26 | 17 | 10
Participants | 0 | 3 | 2 | 0

6. Primary Outcome: Number of Participants With Specific Liver Laboratory Abnormalities
Description: On-treatment laboratory evaluations are evaluations taken after the day (and time, if collected and not missing) of first dose of study treatment. For participants who are off study treatment, evaluations were within a safety window of 30 days after the last dose of study treatment.
  ALT = Alanine Aminotransferase AST = Aspartate Aminotransferase ULN = Upper Limit of Normal.
Time Frame: From first dose to 30 days post last dose of study treatment (an average of 45 weeks up to approximately 64 weeks)
Population: All randomized participants who received at least one dose of any study medication and had at least one on-treatment liver laboratory measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab | Arm B: Nivolumab Plus Intravesical BCG | Arm C: Nivolumab Plus BMS-986205 | Arm D: Nivolumab Plus BMS-986205 Plus Intravesical BCG
Number analyzed (Participants) | 16 | 26 | 17 | 10
Participants
  ALT OR AST > 3XULN | 0 | 1 | 7 | 2
  ALT OR AST> 5XULN | 0 | 0 | 5 | 1
  ALT OR AST> 10XULN | 0 | 0 | 1 | 1
  ALT OR AST > 20XULN | 0 | 0 | 1 | 0
  TOTAL BILIRUBIN > 2XULN | 0 | 0 | 1 | 1
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>1.5XULN IN 1 DAY | 0 | 0 | 1 | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>1.5XULN IN 30 DAYs | 0 | 0 | 1 | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 1 DAY | 0 | 0 | 1 | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 30 DAYS | 0 | 0 | 1 | 0
  ALP>1.5XULN | 0 | 2 | 1 | 0

7. Primary Outcome: Number of Participants With Specific Thyroid Laboratory Abnormalities
Description: On-treatment laboratory evaluations are evaluations taken after the day (and time, if collected and not missing) of first dose of study treatment. For participants who are off study treatment, evaluations were within a safety window of 30 days after the last dose of study treatment.
  TSH = Thyroid Stimulating Hormone LLN = Lower Limit of Normal ULN = Upper Limit of Normal
Time Frame: From first dose to 30 days post last dose of study treatment (an average of 45 weeks up to approximately 64 weeks)
Population: All randomized participants who received at least one dose of any study medication and had at least one on-treatment thyroid laboratory measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab | Arm B: Nivolumab Plus Intravesical BCG | Arm C: Nivolumab Plus BMS-986205 | Arm D: Nivolumab Plus BMS-986205 Plus Intravesical BCG
Number analyzed (Participants) | 16 | 26 | 16 | 10
Participants
  TSH > ULN | 5 | 5 | 2 | 1
  TSH > ULN WITH TSH <= ULN AT BASELINE | 4 | 5 | 1 | 1
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 2 | 1 | 2 | 0
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 2 | 3 | 1 | 0
  TSH > ULN WITH FT3/FT4 TEST MISSING | 2 | 3 | 0 | 1
  TSH < LLN | 2 | 3 | 3 | 1
  TSH <LLN WITH TSH >= LLN AT BASELINE | 2 | 3 | 3 | 1
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 2 | 1 | 1 | 1
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 1 | 3 | 0 | 0
  TSH < LLN WITH FT3/FT4 TEST MISSING | 0 | 0 | 2 | 0

8. Primary Outcome: Number of Participants With Changes From Baseline Laboratory Values
Description: On-study laboratory parameters include hematology, chemistry, liver function, and renal function. On-study laboratory evaluations are evaluations taken after the day (and time, if collected and not missing) of first dose of study treatment. For participants who are off study treatment, evaluations were within a safety window of 30 days after the last dose of study treatment. On-study lab parameters are reported using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: From baseline to 30 days post last dose of study treatment (an average of 45 weeks up to approximately 64 weeks)
Population: All randomized participants who received at least one dose of any study medication and had at least one on-study select laboratory measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab | Arm B: Nivolumab Plus Intravesical BCG | Arm C: Nivolumab Plus BMS-986205 | Arm D: Nivolumab Plus BMS-986205 Plus Intravesical BCG
Number analyzed (Participants) | 16 | 26 | 17 | 10
Participants
  Hemoglobin | 1 | 7 | 5 | 6
  Platelet Count | 1 | 1 | 1 | 1
  Leukocytes, Local Lab | 0 | 0 | 4 | 0
  Lymphocytes (Absolute): number analyzed (Participants) | 2 | 2 | 6 | 0
  Lymphocytes (Absolute) | 0 | 0 | 3 | 0
  Lymphocytes (Absolute), Local Lab: number analyzed (Participants) | 14 | 24 | 11 | 10
  Lymphocytes (Absolute), Local Lab | 2 | 7 | 2 | 5
  Absolute Neutrophil Count | 0 | 1 | 1 | 0
  Alkaline Phosphatase (ALP), Local Lab | 0 | 2 | 2 | 1
  Aspartate Aminotransferase (AST), Local Lab | 3 | 5 | 12 | 3
  Alanine Aminotransferase (ALT), Local Lab | 4 | 10 | 13 | 7
  Bilirubin Total, Local Lab | 1 | 2 | 5 | 3
  Creatinine, Local Lab: number analyzed (Participants) | 16 | 25 | 15 | 10
  Creatinine, Local Lab | 1 | 8 | 3 | 5
  Hypernatremia | 0 | 3 | 4 | 2
  Hyponatremia | 4 | 3 | 4 | 3
  Hyperkalemia | 0 | 3 | 2 | 3
  Hypokalemia | 2 | 2 | 1 | 1
  Hypercalcemia: number analyzed (Participants) | 16 | 26 | 17 | 9
  Hypercalcemia | 2 | 4 | 0 | 3
  Hypocalcemia: number analyzed (Participants) | 16 | 26 | 17 | 9
  Hypocalcemia | 0 | 1 | 2 | 2
  Hypermagnesemia | 3 | 1 | 2 | 0
  Hypomagnesemia | 1 | 3 | 1 | 3
  Hyperglycemia: number analyzed (Participants) | 6 | 8 | 9 | 2
  Hyperglycemia | 4 | 1 | 3 | 1
  Hypoglycemia: number analyzed (Participants) | 14 | 22 | 15 | 6
  Hypoglycemia | 0 | 1 | 1 | 0

9. Primary Outcome: Number of Participants With Adverse Events (AEs) by Anti-Drug- Antibody (ADA) Status
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment.
  An Anti-drug antibody (ADA) is defined as biologic drug-reactive antibody, including pre-existing host antibodies that are cross-reactive with the administered biologic drug.
  An ADA-positive participant has at least one ADA positive-sample relative to baseline at any time after initiation of treatment An ADA-negative participant doesn't not have an ADA-positive sample after the initiation of treatment.
Time Frame: From first dose to 30 days post last dose of study treatment (an average of 45 weeks up to approximately 64 weeks)
Population: All randomized participants who received at least one dose of any study medication and had evaluable ADA status.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab | Arm B: Nivolumab Plus Intravesical BCG | Arm C: Nivolumab Plus BMS-986205 | Arm D: Nivolumab Plus BMS-986205 Plus Intravesical BCG
Number analyzed (Participants) | 11 | 22 | 13 | 9
Participants
  Nivolumab ADA Positive: number analyzed (Participants) | 0 | 1 | 1 | 0
  Nivolumab ADA Positive |  | 1 | 1 |
  Nivolumab ADA Negative: number analyzed (Participants) | 11 | 21 | 12 | 9
  Nivolumab ADA Negative | 11 | 21 | 11 | 9

10. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) by Anti-Drug- Antibody (ADA) Status
Description: Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose:
  * Results in death
  * Is life-threatening (an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe)
  * Requires inpatient hospitalization or causes prolongation of existing hospitalization.
  An Anti-drug antibody (ADA) is defined as biologic drug-reactive antibody, including pre-existing host antibodies that are cross-reactive with the administered biologic drug.
  An ADA-positive participant has at least one ADA positive-sample relative to baseline at any time after initiation of treatment An ADA-negative participant doesn't not have an ADA-positive sample after the initiation of treatment.
Time Frame: From first dose to 30 days post last dose of study treatment (an average of 45 weeks up to approximately 64 weeks)
Population: All randomized participants who received at least one dose of any study medication and had evaluable ADA status.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab | Arm B: Nivolumab Plus Intravesical BCG | Arm C: Nivolumab Plus BMS-986205 | Arm D: Nivolumab Plus BMS-986205 Plus Intravesical BCG
Number analyzed (Participants) | 11 | 22 | 13 | 9
Participants
  Nivolumab ADA Positive: number analyzed (Participants) | 0 | 1 | 1 | 0
  Nivolumab ADA Positive | 0 | 1 | 0 | 0
  Nivolumab ADA Negative: number analyzed (Participants) | 11 | 21 | 12 | 9
  Nivolumab ADA Negative | 1 | 3 | 4 | 4

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from the date of their randomization until study completion (assessed up to approximately 48 months). SAEs and Other AEs were assessed from first dose to 100 days after last dose of study therapy (an average of 45 weeks up to approximately 74 weeks).
Arm/Group | Arm A: Nivolumab | Arm B: Nivolumab Plus Intravesical BCG | Arm C: Nivolumab Plus BMS-986205 | Arm D: Nivolumab Plus BMS-986205 Plus Intravesical BCG
All-Cause Mortality (participants affected / at risk) | 0/16 | 3/26 | 2/17 | 0/10
Serious Adverse Events (participants affected / at risk) | 4/16 | 7/26 | 7/17 | 5/10
Other Adverse Events (participants affected / at risk) | 15/16 | 26/26 | 15/17 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivolumab (N=16) | Arm B: Nivolumab Plus Intravesical BCG (N=26) | Arm C: Nivolumab Plus BMS-986205 (N=17) | Arm D: Nivolumab Plus BMS-986205 Plus Intravesical BCG (N=10)
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 1 | 0 | 0
Disease recurrence (General disorders) | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0
Post procedural sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivolumab (N=16) | Arm B: Nivolumab Plus Intravesical BCG (N=26) | Arm C: Nivolumab Plus BMS-986205 (N=17) | Arm D: Nivolumab Plus BMS-986205 Plus Intravesical BCG (N=10)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Glucocorticoid deficiency (Endocrine disorders) | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 1 | 3 | 2 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1
Metamorphopsia (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 2 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 2 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 4 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 2 | 3
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Asthenia (General disorders) | 1 | 1 | 2 | 2
Chills (General disorders) | 0 | 0 | 0 | 2
Fatigue (General disorders) | 3 | 9 | 3 | 4
Gait disturbance (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 5
Localised oedema (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 2 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 2
Thirst (General disorders) | 0 | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 1
Bacterial disease carrier (Infections and infestations) | 0 | 1 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 2 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0
Groin infection (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 1 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 1
Orchitis (Infections and infestations) | 1 | 0 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 2 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 9 | 2 | 3
Wound infection (Infections and infestations) | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 3
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0
Stoma site hypergranulation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Vascular access site rash (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 4 | 4
Amylase increased (Investigations) | 0 | 0 | 1 | 1
Antinuclear antibody positive (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 5 | 4
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 4
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 1 | 0
Blood methaemoglobin present (Investigations) | 0 | 0 | 0 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 1 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 2 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 1
Carbohydrate antigen 19-9 increased (Investigations) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1 | 0
Heart rate irregular (Investigations) | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1 | 1
Neutrophil count increased (Investigations) | 1 | 0 | 0 | 0
Neutrophil percentage increased (Investigations) | 1 | 0 | 0 | 0
PCO2 increased (Investigations) | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 1 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 6 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 3 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 2 | 1
Persistent depressive disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 2
Bladder spasm (Renal and urinary disorders) | 0 | 3 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 10 | 1 | 4
Haematuria (Renal and urinary disorders) | 4 | 11 | 4 | 5
Hypertonic bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 7 | 0 | 4
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 8 | 1 | 7
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal mass (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 1
Strangury (Renal and urinary disorders) | 0 | 2 | 0 | 0
Urethral pain (Renal and urinary disorders) | 1 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 3 | 1 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 1 | 2
Ejaculation disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 2 | 0 | 0
Testicular mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 6 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
As of early April 2021, Study CA2099UT enrollment was significantly behind the projected target enrollment, (number of participants enrolled 142; target enrollment 480). Since the study would be unable to meet the scientific objectives within a projected timeline, a decision was made in May 2021 to close the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT03519256/Prot_SAP_000.pdf